CLINICAL TRIAL: NCT02703025
Title: CLINICAL EVALUATION OF GCB-70 IN OVERWEIGHT SUBJECTS:An Add-On Study
Brief Title: Evaluation of GCB-70 in Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chemical Resources (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PROTOCOL NO. CR-GCB- 70/ 07/14
Record Dates: First submitted 2015-09-30; First posted 2016-03-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-04

CONDITIONS: Weight Loss
Keywords: Obesity, green coffee bean extract, weight management
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: open level
Oversight: Data Monitoring Committee: No

ARMS (1):
- GCB 70 administered group (Experimental): Green coffee bean extract capsule 500mg, BD
  Interventions: Dietary Supplement: GCB-70

INTERVENTIONS:
Dietary Supplement: GCB-70 — green coffee bean extract

SUMMARY:
Clinical evaluation of GCB-70 in overweight subjects: An Add-On Study

DETAILED DESCRIPTION:
In recent years the prevalence of obesity has increased reaching epidemic levels. Obesity can be defined as excess accumulation of body fat arising from a sustained or a periodic positive energy balance that is when energy intake exceeds energy expenditure. Overweight and obesity is based on Body Mass Index (BMI) Accordingly to the World Health Organization (WHO) classifies individuals with BMI 25-29.99 kg/m2 as overweight while individuals with BMI≥ 30 kg/m2 are termed obese. Apart from being a major contributor to chronic disease burden and mortality, obesity-particularly abdominal obesity, is also closely related to the metabolic syndrome, a cluster of diseases that encompasses the following conditions Dyslipidemia, Hypertension Glucose intolerance and insulin resistance.Abdominal obesity The World Health Organization predicts there will be 2.3 billion overweight adults in the world by 2015, and more than 700 million of them will be obese. Worldwide obesity has more than doubled since 1980. In 2008, 1.5 billion adults, 20 years of age and older, were overweight. Of these, over 200 million men and nearly 300 million women were obese. Over 65% of the world population lives in countries where overweight and obesity kills more people than underweight .

Overweight and obesity have become a serious health concern . Diﬀerent weight management strategies are presently utilized and a variety of weight loss supplements sold as "slimming aids" are readily available. However, the eﬃcacy of some of these food supplements remains uncertain. With the high cost of prescription weight loss drugs and the fear of side effects, the general public is turning to nutraceuticals. One such supplement is the green coﬀee extract (GCE).GCE is present in green or raw coﬀee.

Coffee (Coffea L.) is the world's favourite beverage and the second-most traded commodity after oil. In 2009/10 coffee accounted for exports worth an estimated US$ 15.4 billion, when some 93.4 million bags were shipped, with total coffee sector employment estimated at about 26 million people in 52 producing countries. Arabica coffee (Coffea arabica L.) and robusta coffee (C. canephora Pierre ex A.Froehner) are the two main species used in the production of coffee. 66% of the world production mostly comes from Coffea arabica L. and 34% from Coffea canephora. Coffee belongs to family Rubiaceae in the genus Coffea.

GCB-70 is obtained from raw seeds or beans of Coffee. In producing the normal coffee for sale, the berries are roasted to produce the traditional beverage. However, no roasting is done for green extract so as to preserve important components

ELIGIBILITY:
Inclusion Criteria:

1. Agrees to written as well as audio-visual informed consent
2. Patients of either sex.
3. BMI >25 kg/m2
4. Aged 18-65 years
5. Euthyroid
6. Not receiving any steroids

Exclusion Criteria:

i. Uncooperative Subjects ii. Lactating and Pregnant or planning to conceive females. iii. Physically/ mentally unwell as certified by physician-in-charge. iv. Participation in any other clinical trial with in the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Narsingh Verma, MD, Principal Investigator — Dept of Physiology,King George's Medical University, Lucknow, UP, India
Locations (1):
- Department of Physiology, King George's Medical University, Lucknow, UP, India, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No